CLINICAL TRIAL: NCT04786431
Title: Shotgun Mass Spectrometry-based Lipid Profiling in Chronic Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Hospital Santa Cruz, Centro Hospitalar de Lisboa Ocidental (Unknown); Department of Neurology, Hospital de Egas Moniz, Centro Hospitalar de Lisboa Ocidental (Unknown); Hospital Dr. Fernando da Fonseca (Unknown); Lipotype GmbH, Tatzberg 47, 01307, Dresden, Germany. (Unknown); iNOVA4Health, CEDOC, NOVA Medical Schoo (Unknown); Fundação para a Ciência e a Tecnologia (FCT) (Unknown)
Responsible Party: Sponsor
Other Study IDs: UniversidadeNL_29395
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Biomarker; Lipid; Inflammation; Cardiovascular Diseases; Ischemic Stroke; Systemic Lupus Erythematosus; Healthy
Keywords: Mass spectromtry; Lipidomics; cardiovascular disease; Machine learning; Regression models
MeSH Terms: conditions — Inflammation; Cardiovascular Diseases; Ischemic Stroke; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples were drawn into tubes containing an anti-coagulant (heparin or EDTA) immediately after admission into the hospital and signing of the informed consent. The samples were kept at 4°C and processed within 24 h from collection. Plasma was obtained by centrifugation of the blood at 500 g for 10 min at 4°C, frozen at -80°C and stored at this temperature until they were used for the lipidomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Controls, CVD, IS, SLE: Control (n = 85) were taken from the population of the Coimbra and Lisbon, Portugal, regions. They satisfied the criterion that they had never had any CVD- or SLE-related health complaints.
  The CVD patients (n = 238) were divided into 6 groups. CVD1 (n = 61) contains individuals who went to the hospital with chest pain but had no indicators for stable angina pectoris, unstable angina pectoris or myocardial infarction.
  Acute ischemic stroke (IS) (n = 21) were patients admitted at the emergency room of the Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal, who suffered from acute ischemic stroke.
  The SLE cohort (n = 104) were patients from Hospital Dr. Fernando Fonseca, Amadora, Portugal.
  Interventions: Other: Blood collection for lipid profiling by LC-MS

INTERVENTIONS:
Other: Blood collection for lipid profiling by LC-MS — Blood withdrawal

SUMMARY:
Collect blood from patients admitted for coronary angiography to tubes with heparin, centrifuge and collect plasma. This will be frozen at -80C. Sent to the Lipotype laboratory, Dresden, Germany, for the detection and quantification of compounds derived from oxidized LDL cholesterol (cholesterol hemi-esters).

DETAILED DESCRIPTION:
Plasma samples were obtained from a total of 427 individuals. Baseline characteristics are outlined in Table 1. Control (n = 85) were taken from the population of the Coimbra and Lisbon, Portugal, regions. They satisfied the criterion that they had never had any CVD- or SLE-related health complaints. The CVD patients (n = 238) were divided into 6 groups. CVD1 (n = 61) contains individuals who went to the hospital with chest pain but had no indicators for stable angina pectoris, unstable angina pectoris or myocardial infarction. CVD2 (n = 82) are patients with stable angina pectoris (SAP). CVD1 and CVD2 are defined according to the ACCF/AHA/ACP/AATS/PCNA/SCAI/STS guidelines. CVD3 (n = 20) contains patients with unstable angina pectoris, CVD4 (n = 34) are patients who suffered an acute myocardial infarction with no ST-elevation in ECG, and CVD5 (n = 20) are patients who suffered acute myocardial infarction with ST-elevation in ECG. CVD3, CVD4, and CVD5, together, may be classified as patients with an acute coronary syndrome (ACS). CVD1 through CVD5 groups were all obtained from Hospital Santa Cruz, Carnaxide, Portugal. Acute ischemic stroke (IS) (n = 21) were patients admitted at the emergency room of the Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal, who suffered from acute ischemic stroke. The SLE cohort (n = 104) were patients from Hospital Dr. Fernando Fonseca, Amadora, Portugal. The inclusion criteria were all patients diagnosed with the pathology and above 18 years old. The exclusion criteria were the existence of serious renal and hepatic pathologies, cancer or existence of infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for coronary angiography due to suspected coronary disease (silent ischemia, stable angina and acute coronary syndromes)

Exclusion Criteria:

* Patients unable to give informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Controls were from the population of the Coimbra and Lisbon, Portugal, regions. They satisfied the criterion that they had never had any CVD- or SLE-related health complaints. CVD1 (n= 61) contains individuals who went to the hospital with chest pain but had no indicators for stable angina pectoris, unstable angina pectoris or myocardial infarction. CVD2 (n=82) are patients with stable angina pectoris. CVD3 (n=20) contains patients with unstable angina pectoris, CVD4 (n=34) are patients who suffered an acute myocardial infarction with no ST-elevation in ECG, and CVD5 (n= 20) are patients who suffered acute myocardial infarction with ST-elevation in ECG. CVD1 through CVD5 groups were from Hospital Santa Cruz, Carnaxide, Portugal. IS (n=21) were patients admitted at the emergency room of the Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal, who suffered from acute ischemic stroke. The SLE cohort (n=104) were patients from Hospital Dr. Fernando Fonseca, Amadora, Portugal.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of inflammatory disease | Day 1: Age, height, weight, sex, statin use and lipid level in plasma
  Controls never had any CVD- or SLE-related health complaints.
  CVD1 contains individuals who went to the hospital with chest pain but had no indicators for stable angina pectoris, unstable angina pectoris or myocardial infarction. CVD2 are patients with stable angina pectoris (SAP). CVD1 and CVD2 are defined according to the ACCF/AHA/ACP/AATS/PCNA/SCAI/STS guidelines. CVD3 contains patients with unstable angina pectoris, CVD4 are patients who suffered an acute myocardial infarction with no ST-elevation in ECG, and CVD5 are patients who suffered acute myocardial infarction with ST-elevation in ECG .
  Acute ischemic stroke (IS) were patients admitted at the emergency room of the Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal
  SLE cohort were patients from Hospital Dr. Fernando Fonseca, Amadora, Portugal.

CONTACTS AND LOCATIONS:
Overall Officials: Otília Vieira, PhD, Principal Investigator — iNOVA4Health, CEDOC, NOVA Medical School, NMS, Universidade Nova de Lisboa, 1169-056 Lisboa, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fihn SD, Gardin JM, Abrams J, Berra K, Blankenship JC, Dallas AP, Douglas PS, Foody JM, Gerber TC, Hinderliter AL, King SB 3rd, Kligfield PD, Krumholz HM, Kwong RY, Lim MJ, Linderbaum JA, Mack MJ, Munger MA, Prager RL, Sabik JF, Shaw LJ, Sikkema JD, Smith CR Jr, Smith SC Jr, Spertus JA, Williams SV. 2012 ACCF/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the Diagnosis and Management of Patients With Stable Ischemic Heart Disease: Executive Summary: A Report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines, and the American College of Physicians, American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2012 Dec 18;60(24):2564-603. doi: 10.1016/j.jacc.2012.07.012. Epub 2012 Nov 19. No abstract available. PMID 23182124
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members; Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):2354-94. doi: 10.1161/CIR.0000000000000133. Epub 2014 Sep 23. No abstract available. PMID 25249586